CLINICAL TRIAL: NCT05818618
Title: Impact of Topical Clobetasol on Gingival Crevicular Fluid miRNAs in Subjects Affected by Oral Lichen Planus: a Randomized Clinical Trial
Brief Title: Impact of Topical Clobetasol on Gingival Crevicular Fluid miRNAs in Subjects Affected by Oral Lichen Planus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Catania (Other)
Responsible Party: Principal Investigator, Gaetano Isola, Researcher, University of Catania
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 121-21
Record Dates: First submitted 2023-04-05; First posted 2023-04-19 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Oral Lichen Planus
MeSH Terms: conditions — Lichen Planus, Oral

STUDY DESIGN:
Intervention Model Description: The main aim of the study is to analyze the impact of topical clobetasol on gingival crevicular fluid miRNAs expression in subjects affected by oral lichen planus.
Who Masked: Participant, Investigator
Masking Description: Sealed envelopes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clobetasol propionate 0,05% gel (Active Comparator): Patients were treated with a topic gel of clobetasol propionate 0,05%
  Interventions: Drug: Clobetasol Topical Gel
- Placebo (Placebo Comparator): Patients were treated with a topic placebo gel control
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Clobetasol Topical Gel — Topic Clobetasol gel applied locally on OLP lesions.
  Arms: Clobetasol propionate 0,05% gel
Drug: Placebo — Placebo oral gel applied locally on OLP lesions.
  Arms: Placebo

SUMMARY:
According to recent research, microRNAs (miRNAs) may function as early disease indicators and contribute to the severity of a number of precancerous and malignant oral disorders. The aim of the present study, through a double-blind randomized controlled trial design, is to analyze in the gingival crevicular fluid (GCF) as a non-invasive approach the impact of topical clobetasol on miRNAs expression in subjects affected by oral lichen planus (OLP).

DETAILED DESCRIPTION:
A double-blind randomized controlled clinical trial is conducted in order to evaluate the impact of topical clobetasol on GCF miRNAs expression in subjects with OLP and determine the statistical significance of the outcome variables.

At least 60 patients with OLP, randomly allocated in two groups: placebo group with a 4% hydroxyethyl cellulose adhesive gel and the clobetasol group with the same gel containing clobetasol propionate 0,05%.

ELIGIBILITY:
Inclusion Criteria:

* The complete correspondence of the most recent WHO clinical and histopathological criteria (2020) for OLP diagnosis.

Exclusion Criteria:

* 1) Previous therapies for OLP during the last six months preceding the study; 2) State of pregnancy or breastfeeding; 3) Contact or drug oral lichenoid lesions; 4) Allergies to the molecules used in the study; 5) HIV seropositivity.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2020-03-12 (Actual); Primary Completion 2023-07-05 (Actual); Study Completion 2023-08-10 (Actual)

PRIMARY OUTCOMES:
miRNAs GCF levels | 8 weeks
  The level of expression of different miRNAs in the GCF before and after treatment in the two groups. (Scale 0-4)

SECONDARY OUTCOMES:
OLP disease severity scores | 8 weeks
  The eventual improvement in OLP symptoms, signs and disease severity scores after treatment in the two groups. (Scale 0-4)

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano Isola, Principal Investigator — University of Catania
Locations (1):
- AOU Policlinico G. Rodolico, Catania, Italy

IPD SHARING:
Plan to Share IPD: Yes
Study protocol
Time Frame: 5 months
Access Criteria: Pubmed